CLINICAL TRIAL: NCT03368248
Title: Evaluation of the Palliative Approach in the NICU
Acronym: EvDPMNN
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD1415
Record Dates: First submitted 2017-11-24; First posted 2017-12-11 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Neonatal Death
Keywords: Palliative care; Collegial meetings; Neonatal resuscitation services; Survey; Medico-caring staff of the NICUs
MeSH Terms: conditions — Perinatal Death | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All neonatal resuscitation services.: All professionals in contact with children were interviewed: doctors (senior and intern), paramedics (managers, pediatric nurses, auxiliaries and nurses, psychomotor therapists) and psychologists. The survey was based on a questionnaire, which was offered to all professionals, both medical and non-medical.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — A survey was conducted among all professionals in neonatal resuscitation services : doctors (senior and intern), paramedics (managers, pediatric nurses, auxiliaries and nurses, psychomotor therapists) and psychologists. The survey was based on a questionnaire, which was offered to all professionals, both medical and non-medical. All questions were closed, and a free comment area was proposed at the end. The questionnaire was preceded by a comment recalling the objectives of the study, the voluntary and individual nature of participation, and insisted on respect for anonymity. It consisted of 49 questions, allowing 197 possible answers. For most questions, several answers could be chosen.

SUMMARY:
In neonatal resuscitation, the majority of deaths currently occur after a Life Limitation or Discontinuance (LAT) procedure. In the 1990s, the approach was different, as Marina CUTTINI put it in a European study that highlighted some French peculiarities: doctors and nurses found it legitimate to have life stops in certain circumstances, and wanted to keep parents away from these decisions deemed guilt. Civil society has changed the thinking in recent years by the so-called Kouchner then LEONETTI laws. The palliative approach, which is defined as the search for a fair and reasonable balance, constantly reevaluated, between curative care and care of comfort and support, has become a constant concern in neonatal resuscitation services. However, we did not find a recent study that specifies in France the modalities of deaths in neonatology, especially their proportion after LAT. Also, shortly before the adoption of the CLAYES-LEONETTI law, the authors wished to make an inventory of the practices of all the neonatal intensive care units of Ile de France, one of the main centers of French fertility.

The objectives of the study were to describe the organization of collegial meetings (CR), the decision-making process and implementation of LATs, with particular attention to stopping artificial nutrition and hydration, and sedation / analgesia. The place of the parents in these different processes (gathering their opinion, information on how to withdraw life-saving treatment, leading in the event of disagreement) was also studied. Finally, some questions about euthanasia were asked, in order to measure the evolution of ideas and practices more than 15 years after EURONIC and 10 years after the LEONETTI law.

DETAILED DESCRIPTION:
This is a survey carried out among all neonatal resuscitation services in the Ile-de-France region, from January 1 to 31, 2016. All professionals in contact with children were interviewed: doctors (senior and intern), paramedics (managers, pediatric nurses, auxiliaries and nurses, psychomotor therapists) and psychologists. The survey was based on a questionnaire, which was offered to all professionals, both medical and non-medical. All questions were closed, and a free comment area was proposed at the end. The questionnaire was preceded by a comment recalling the objectives of the study, the voluntary and individual nature of participation, and insisted on respect for anonymity. It consisted of 49 questions, allowing 197 possible answers. For most questions, several answers could be chosen. An additional questionnaire was sent to the heads of the services, medical and care settings. The questions sought to describe the 2014 activity (number of admissions and number of deaths, number of collegiate meetings and number of deaths resulting from an LAT), medical and paramedical staff to calculate the response rate, the existence of reflection and / or training on palliative and end-of-life care in the service, as well as the existence of a mobile team or palliative care unit in the facility.

ELIGIBILITY:
Inclusion Criteria:

* medico-caring staff of the NICUs in the Paris region

Exclusion Criteria:

* No response to the supplementary questionnaire, not allowing to assess the response rate of the center

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Medico-caring staff of the NICUs in the Paris region.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-04-01 (Actual)

PRIMARY OUTCOMES:
Measure the level of appropriation by neonatal resuscitation services in the Paris region of the legal devices related to the palliative approach. | Through study completion, an average of four months.
  The questions were designed to measure the level of training of medical and paramedical personnel on palliative and end-of-life care in the service.

SECONDARY OUTCOMES:
Measure the level of each death patterns in neonatal resuscitation services in the Paris region. | Through study completion, an average of four months.
  To measure the implementation of the limitations and shutdowns of active therapies, with particular attention to stopping artificial nutrition and hydration, as well as stopping sedation. To measure precisely this data it will be necessary to answer the questionnaire of the study. Questions about death patterns will account for the number of deaths associated with an interruption of artificial nutrition, a cessation of hydration or cessation of sedation. This will allow the data to be encrypted for use.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BOIZE, Principal Investigator — Hôpital NOVO

IPD SHARING:
Plan to Share IPD: No